CLINICAL TRIAL: NCT03974308
Title: Effectiveness of Spa Treatment in Patients With Spine Osteoarthritis in Comparison With Outpatient Physiotherapy and no Physiotherapy
Brief Title: Effectiveness of Spa Treatment, Outpatient Physiotherapy and no Physiotherapy in Spine Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Jolanta Zwolińska, Head of the Laboratory of Physical Factors, University of Rzeszow
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Spa treatment
Record Dates: First submitted 2018-05-11; First posted 2019-06-04 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Spine Osteoarthritis; Spa Resorts
Keywords: Balneotherapy; Health Resorts; Quality of life
MeSH Terms: conditions — Osteoarthritis, Spine | interventions — Balneology

STUDY DESIGN:
Intervention Model Description: Comparison of the level of pain, life satisfaction and level of disability in people with degenerative spine disease which:
  1. use the spa treatment
  2. use complex physiotherapy in the place of residence
  3. don't use physiotherapy, ad hoc pharmacotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group 1 (Experimental): Patients with spine osteoarthritis who will be treated in polish spas in Subcarpathian Region. Comprehensive physiotherapy including balneotherapy will be applied.
  Interventions: Other: Comprehensive physiotherapy including balneotherapy and filling questionaire
- Study group 2 (Active Comparator): Patients with spine osteoarthritis who will be treated in outpatient treatment. Comprehensive physiotherapy without balneotherapy will be applied.
  Interventions: Other: Comprehensive physiotherapy without balneotherapy and filling questionaire
- Control group (Other): Patients with spine osteoarthritis who will not have applied physiotherapy nor balneotherapy.
  Interventions: Other: No intervention, only filling questionaire

INTERVENTIONS:
Other: Comprehensive physiotherapy including balneotherapy and filling questionaire — Three-week stay in a sanatorium with comprehensive physiotherapy including balneotherapy and three time filling questionaire.
  Other Names: Sanatorium treatment
  Arms: Study group 1
Other: Comprehensive physiotherapy without balneotherapy and filling questionaire — Two-week outpatient treatment with comprehensive physiotherapy without balneotherapy and three time filling questionaire
  Other Names: Outpatient physiotherapy
  Arms: Study group 2
Other: No intervention, only filling questionaire — No physiotherapy nor balneotherapy applied but three time filling questionaire
  Arms: Control group

SUMMARY:
In the first study group will participate patients with spine osteoarthritis who will be treated in polish spas in Subcarpathian Region. Complex physiotherapy including balneotherapy will be applied in study group participants. In the second study group will participate patients with spine osteoarthritis who will be treated in outpatient treatment. Complex physiotherapy without balneotherapy will be applied in second study group participants. In the control group will participate patients with spine osteoarthritis who will not have applied physiotherapy nor balneotherapy during observation. In all patients will be evaluated quality of life, level of pain intensity and health assessment.

DETAILED DESCRIPTION:
The following questionnaires will be used: original socio-demographic data questionnaire, the VAS (visual analogue scale) pain severity rating scale, the modified Laitinen pain questionnaire, the Life Satisfaction Questionnaire LISAT-9 and the HAQ: Health Assesment Questionnaire.

Questionnaires will be completed: before the beginning of therapy, one month and six months after the end of therapy.

Questionnaires in control group will be completed: in the beginning of observation and in the same time intervals as in study groups.

ELIGIBILITY:
Inclusion Criteria:

* Spine osteoarthritis

Exclusion Criteria:

* no consent to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Health Assesment Questionaire (HAQ) | Change from baseline HAQ value at month and six months after therapy
  Subjective assesment of level of disability. Value of each of 8 subsections: minimum value 0, maximum value 3. total score is averaged. the best total score is 0, the worst is 3.

SECONDARY OUTCOMES:
Laitinen Pain Indicator Questionnaire | Change from baseline Laitinen value at month and six months after therapy
  pain severity rating scale. Each subsection is considered separately and total score is considered summed. In each of 4 subsections minimum value is 0, maximum value is 4. the best score is 0, the worst is 4.
Visual Analogue Scale (VAS) | Change from baseline VAS value at month and six months after therapy
  pain severity rating scale. only one value. Minimium value is 0, maximum value is 10. the best is 0, the worst is 10.

OTHER OUTCOMES:
Life Satisfaction Questionnaire (LISAT-9) | Change from baseline LISAT-9 value at month and six months after therapy
  Subjective assesment of life satisfaction. Each of 9 subsections is considered separately and in total. Minimum value in each subsection is 1, maximum value is 6. Total score is averaged. The best value is 6, the worst is 1.

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Zwolińska, PhD, Principal Investigator — University of Rzeszow
Locations (1):
- University of Rzeszow, Rzeszów, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karagulle M, Karagulle MZ. Effectiveness of balneotherapy and spa therapy for the treatment of chronic low back pain: a review on latest evidence. Clin Rheumatol. 2015 Feb;34(2):207-14. doi: 10.1007/s10067-014-2845-2. Epub 2014 Dec 23. PMID 25535198
- [Background] Verhagen A, Bierma-Zeinstra S, Lambeck J, Cardoso JR, de Bie R, Boers M, de Vet HC. Balneotherapy for osteoarthritis. A cochrane review. J Rheumatol. 2008 Jun;35(6):1118-23. Epub 2008 May 1. PMID 18464302
- [Background] Fortunati NA, Fioravanti A, Seri G, Cinelli S, Tenti S. May spa therapy be a valid opportunity to treat hand osteoarthritis? A review of clinical trials and mechanisms of action. Int J Biometeorol. 2016 Jan;60(1):1-8. doi: 10.1007/s00484-015-1030-x. Epub 2015 Jul 9. PMID 26156832
- [Result] Mordarski S. Pain management in the elderly: transdermal fentanyl for the treatment of pain caused by osteoarthritis of the knee and hip. Biomed Res Int. 2014;2014:262961. doi: 10.1155/2014/262961. Epub 2014 Jan 5. PMID 24527441
- [Result] Li Y, Wei X, Zhou J, Wei L. The age-related changes in cartilage and osteoarthritis. Biomed Res Int. 2013;2013:916530. doi: 10.1155/2013/916530. Epub 2013 Jul 22. PMID 23971049
- [Result] Moskowitz RW. The burden of osteoarthritis: clinical and quality-of-life issues. Am J Manag Care. 2009 Sep;15(8 Suppl):S223-9. PMID 19817508
- [Result] Brown R, Tomasello L, Mitchell DA, Sebald A, Stepney S. Ternary graph as a questionnaire: a new approach to assessment of quality of life? Br J Oral Maxillofac Surg. 2017 Sep;55(7):679-684. doi: 10.1016/j.bjoms.2017.04.011. Epub 2017 May 18. PMID 28528676
- [Result] Lourenco S, Lucas R, Araujo F, Bogas M, Santos RA, Barros H. Osteoarthritis medical labelling and health-related quality of life in the general population. Health Qual Life Outcomes. 2014 Nov 30;12:146. doi: 10.1186/s12955-014-0146-8. PMID 25433808
- [Result] Bellometti S, Gallotti C, Pacileo G, Rota A, Tenconi MT. Evaluation of outcomes in SPA-treated osteoarthrosic patients. J Prev Med Hyg. 2007 Mar;48(1):1-4. PMID 17506230
- [Result] Dandinoglu T, Dandin O, Ergin T, Tihan D, Akpak YK, Aydin OU, Teomete U. Can balneotherapy improve the bowel motility in chronically constipated middle-aged and elderly patients? Int J Biometeorol. 2017 Jun;61(6):1139-1148. doi: 10.1007/s00484-016-1295-8. Epub 2016 Dec 23. PMID 28011998
- [Derived] Zwolinska J, Gasior M. Effects of complex spa therapy in patients with osteoarthritis of the spine receiving treatments in health resorts in south-eastern Poland. Sci Rep. 2022 Aug 29;12(1):14663. doi: 10.1038/s41598-022-18046-6. PMID 36038633